CLINICAL TRIAL: NCT00471835
Title: A Phase I/II Study of Hypofractionated Stereotactic Body Radiotherapy for Stage I/II Non-small Cell Lung Cancer Within the Central Lung Region and the Prognostic Impact of FDG Positron Emission Tomography
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Stage I or Stage II Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CCCWFU-62206; CDR0000543743 (Registry Identifier: PDQ (Physician Data Query)); CCCWFU-IRB00000578
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage I non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Magnetic Resonance Spectroscopy; Radiosurgery

INTERVENTIONS:
Procedure: computed tomography
Procedure: positron emission tomography
Radiation: stereotactic body radiation therapy

SUMMARY:
RATIONALE: Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I/II trial is studying the side effects and best dose of stereotactic body radiation therapy and to see how well it works in treating patients with stage I or stage II non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of hypofractionated stereotactic body radiotherapy (SBRT) to the central lung region (peri-mediastinum) in patients with stage I or II non-small cell lung cancer. (Phase I)
* Determine local control and time to local progression in patients treated with this regimen. (Phase II)
* Evaluate the ability of peak standardized uptake values (SUV) for fludeoxyglucose F 18 (FDG)-PET scan, obtained shortly after SBRT (post-treatment), to predict local control and time to progression in these patients.

Secondary

* Evaluate the ability of maximum SUV for FDG-PET scan, obtained shortly after SBRT, to predict long-term local control and time to progression in these patients.
* Evaluate the ability of peak SUV and max SUV for FDG-PET scan, obtained prior to SBRT, to predict local control and time to progression in these patients.
* Determine the utility of PET/CT scan data in guiding treatment planning.
* Determine if treatment with radiotherapy involving high biological doses with limited treatment volume using these SBRT techniques achieves acceptable treatment-related toxicity.

OUTLINE: This is a phase I dose-escalation study followed by a phase II open-label study.

* Phase I: Patients undergo hypofractionated stereotactic body radiotherapy (SBRT) 3 times within a 2-week time frame.

Cohorts of 3-6 patients receive escalating doses of hypofractionated SBRT until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients undergo hypofractionated SBRT at the MTD as in phase I. In both phases, patients undergo fludeoxyglucose F 18-PET/CT scans at baseline and at 12-16 weeks after completion of SBRT.

After completion of study treatment, patients are followed periodically for 4 years.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage I or II non-small cell lung cancer meeting the following criteria:

  * No bronchoalveolar cell carcinoma
  * Maximum T2 or T3 tumor size ≤ 5 cm

    * T3 primary tumor must be limited to chest wall
  * Primary tumor of any T stage must be within or touching the zone of the trachea or proximal bronchial tree, defined as a volume of 2 cm in all directions around the trachea and proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchi, right middle lobe bronchus, right and left lower lobe bronchi)

    * For lesions inferior to the proximal bronchial tree, the primary tumor must be within 2 cm of the esophagus
  * Patients with N1 (hilar) lymph nodes positive for malignancy based on size, fludeoxyglucose F 18 (FDG)-PET scan uptake, or biopsy are eligible if the N1 lymph nodes are located such that they are contiguously within the same stereotactic radiation treatment field as the primary tumor
  * Mediastinal lymph nodes must be ≤ 1 cm and no abnormal uptake on FDG-PET scan in those areas

    * Patients with > 1 cm lymph nodes or abnormal FDG-PET scan (including suspicious but non-diagnostic uptake) are eligible if directed tissue biopsy of all abnormally identified areas are negative for cancer
* No evidence of distant metastases

  * Suspected M1 disease based on pre-treatment PET imaging must be biopsied

    * If the biopsy is positive, the patient is ineligible
    * If the biopsy is negative and representative of the lesion in question, the patient is eligible
    * If the biopsy is non-diagnostic, consideration should be given to repeat biopsy

      * If the repeat biopsy remains non-diagnostic or a biopsy is not feasible, then the patient is ineligible
* Technically resectable disease

  * Surgery refused or patient deemed medically inoperable due to co-morbid conditions

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No synchronous primary or invasive malignancy within the past 2 years other than non-melanomatous skin cancer
* No active systemic, pulmonary, or pericardial infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chest radiotherapy (lung or mediastinum)
* No other concurrent anticancer therapy, including other radiotherapy, radiofrequency ablation (or other antineoplastic interventional radiology techniques), chemotherapy, biological therapy, vaccine therapy, or surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Maximum tolerated dose (Phase I)
Time to progression and local control at 1 and 2 years (Phase II)

SECONDARY OUTCOMES:
Rate of acute and late treatment-related toxicity related to specific symptoms, including gastrointestinal, cardiac, neurologic, hemorrhagic, and pulmonary symptoms
Toxicity
Patterns of failure and overall survival at 2 years
Measurement of pre-treatment and post-treatment PET scan standardized uptake values and correlation of this data with local control at 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Volker W. Stieber, MD, Study Chair — Wake Forest University Health Sciences